CLINICAL TRIAL: NCT04091282
Title: Antibiotic-induced Disruption of the Maternal and Infant Microbiota and Adverse Health Outcomes - The ABERRANT Study
Brief Title: Antibiotic-induced Disruption of the Microbiota
Acronym: ABERRANT
Status: Recruiting | Type: Observational
Sponsor: University of Fribourg (Other)
Responsible Party: Principal Investigator, Petra Zimmermann, Principal investigator, University of Fribourg
Other Study IDs: 2019 - 01567
Record Dates: First submitted 2019-08-28; First posted 2019-09-16 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Microbiota; Antibiotic Disruption
Keywords: Metagenome; Infants

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Stool, oral swabs, breast milk, blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The use of antibiotics causes profound changes in the microbiota. However, the magnitude of the effect of intrapartum and early-life antibiotics on the breast milk and the infant oral and intestinal microbiota, and whether effects are only short-term or persist long-term remain uncertain and will be determined in this study.

DETAILED DESCRIPTION:
In this prospective cohort study, the investigators will determine the effect of (i) intrapartum antibiotics on the composition of the breast milk, and the infant oral and intestinal microbiota and antibiotic exposure in the first year of life on the composition of the infant intestinal microbiota (including the development and persistence of antibiotic resistance) and (ii) the association of this disruption with adverse health outcomes. (iii) The investigators will also determine the association between the maternal intestinal microbiota, the breast milk microbiota and the infant oral and intestinal microbiota.

ELIGIBILITY:
Inclusion Criteria:

* healthy infants
* term infants (> 37 weeks of gestation)

Exclusion Criteria:

* maternal HIV infection
* maternal hepatitis B or C infection
* antibiotics in the third trimester of pregnancy
* intake of probiotics during pregnancy
* infants with the low birth weight <2500 g
* infants with congenital abnormality

Ages: 1 Day to 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Women who give birth at the Hôpital fribourgeois (HFR) in Fribourg, Switzerland and their infants.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2020-01-25 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Antibiotic-induced disruption of breast milk microbiota | 2 years
  Composition of breast milk microbiota at birth and when infants are 7 days, 1, 2, 4, 6, 12 and 24 months of age.
Antibiotic-Induced disruption the infant stool microbiota | 2 years
  Composition of infant intestinal microbiota at birth and when infants are 7 days, 1, 2, 4, 6, 12 and 24 months of age.
Maternal to infant microbiota transfer | 2 years
  Similarities in the composition of the maternal intestinal, the breast milk microbiota and the infant intestinal microbiota, at 38 weeks of pregnancy, at birth and when infants are 7 days, 1, 2, 4 and 6 months of age.
The composition of the intestinal microbiota and adverse health outcomes | 2 years
  Abundance of certain microbes in the intestinal microbiota and number of episodes of lower respiratory tract infections until 2 years of age
The composition of the intestinal microbiota and adverse health outcomes | 2 years
  Abundance of certain microbes in the intestinal microbiota and number of episodes of acute otitis media episodes until 2 years of age
The composition of the intestinal microbiota and adverse health outcomes | 2 years
  Abundance of certain microbes in the intestinal microbiota and prevalence of allergic sensitisation (positive skin prick test) at 1 and 2 years of age
The composition of the intestinal microbiota and adverse health outcomes | 2 years
  Abundance of certain microbes in the intestinal microbiota and weight (in kg) at 1 and 2 years of age

SECONDARY OUTCOMES:
Antibiotic-induced disruption of breast milk microbiota | 2 years
  Prevalence of antibiotic resistance genes within the breast milk microbiota at birth and when infants are 7 days, 1, 2, 4, 6, 12 and 24 months of age.
Antibiotic-Induced disruption the infant stool microbiota | 2 years
  Prevalence of antibiotic resistance genes within the intestinal microbiota at birth and when infants are 7 days, 1, 2, 4, 6, 12 and 24 months of age.
Introduction of different foods affects the composition of the intestinal microbiota | 2 years
  Age (in days) when a new food item was introduced and composition of infant intestinal microbiota when infants are 1, 2, 4, 6, 12 and 24 months of age.
Administration of oxygen affects the composition of the intestinal microbiota in infants | 2 years
  Number of days of oxygen and composition of infant intestinal microbiota when infants are 7 days, 1, 2, 4, 6, 12 and 24 months of age.
Administration of antacids affect the composition of the infant intestinal microbiota | 2 years
  Number of days antacids were administered and composition of infant intestinal microbiota at birth and when infants are 7 days, 1, 2, 4, 6, 12 and 24 months of age.

CONTACTS AND LOCATIONS:
Overall Officials: Petra Zimmermann, MD, PhD, Principal Investigator — Hopital Cantonal de Fribourg, Switzerland
Locations (1):
- Hopital cantonal Fribourg, Fribourg, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Volery M, Scherz V, Jakob W, Bandeira D, Deggim-Messmer V, Lauber-Biason A, Wildhaber J, Falquet L, Curtis N, Zimmermann P. Study protocol for the ABERRANT study: antibiotic-induced disruption of the maternal and infant microbiome and adverse health outcomes - a prospective cohort study among children born at term. BMJ Open. 2020 Jun 23;10(6):e036275. doi: 10.1136/bmjopen-2019-036275. PMID 32580987